CLINICAL TRIAL: NCT01628601
Title: GANfort® in Patients With Primary Open Angle Glaucoma or Ocular Hypertension Who Are Insufficiently Responsive to Monotherapy
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/027
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Timolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POAG or OHT: Patients with POAG or OHT prescribed GANfort® (fixed combination 0.3 mg bimatoprost and 5 mg timolol) treatment in a dose determined by the physician prior to study entry
  Interventions: Drug: Fixed combination 0.3 mg bimatoprost and 5 mg timolol

INTERVENTIONS:
Drug: Fixed combination 0.3 mg bimatoprost and 5 mg timolol — Patients with POAG or OHT prescribed GANfort® (fixed combination 0.3 mg bimatoprost and 5 mg timolol) treatment in a dose determined by the physician prior to study entry

SUMMARY:
This is an observational study of patients diagnosed with Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT) who are insufficiently responsive to monotherapy and who are prescribed GANfort® (fixed combination of 0.3 mg bimatoprost and 5 mg timolol) by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma or ocular hypertension
* Prescribed GANfort® (fixed combination 0.3 mg bimatoprost and 5 mg timolol)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary open angle glaucoma or ocular hypertension prescribed GANfort® (fixed combination 0.3 mg bimatoprost and 5 mg timolol) by the physician prior to study entry
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | POAG or OHT
Started | 392
Completed | 351
Not Completed | 41

BASELINE CHARACTERISTICS:
Arm/Group | POAG or OHT
Number analyzed (Participants) | 392
Age Continuous [Mean (Standard Deviation); unit: Years] | 67.22 (13.14)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 232
  Male | 155
  Missing Data | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. A negative change from baseline indicates an improvement.
Time Frame: Baseline, 18 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Median (Inter-Quartile Range); unit: Millimeters of Mercury (mmHg)
Arm/Group | POAG or OHT
Number analyzed (Participants) | 345
Millimeters of Mercury (mmHg)
  Baseline - Right Eye (N=345) | 22.0 [18.0 to 24.0]
  Change from Baseline at 18 Wks-Rt Eye (N=345) | -6.0 [-7.0 to -3.0]
  Baseline - Left Eye (N=344) | 22.0 [19.0 to 25.0]
  Change from Baseline at 18 Wks-Lft Eye (N=344) | -6.0 [-7.0 to -4.0]

2. Secondary Outcome: Physician Assessment of Tolerability Using a 4-Point Scale
Description: Physician assessment of tolerability using a 4-point scale (very good, good, moderate, and poor). The number of patients assessed as good and very good combined are reported.
Time Frame: 18 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Number; unit: Participants
Arm/Group | POAG or OHT
Number analyzed (Participants) | 356
Participants | 340

3. Secondary Outcome: Patient Assessment of Tolerability Using a 4-Point Scale
Description: Patient assessment of tolerability using a 4-point scale (very good, good, moderate, and poor). The number of patients assessed as good and very good combined are reported.
Time Frame: 18 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Number; unit: Participants
Arm/Group | POAG or OHT
Number analyzed (Participants) | 349
Participants | 319

4. Secondary Outcome: Physician Assessment of Adherence to GANfort®
Description: Physician Assessment of Adherence to GANfort® was assessed on a 3-point scale (better, equal, and worse). The number of patients assessed as "better" compliance are reported.
Time Frame: 18 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Number; unit: Participants
Arm/Group | POAG or OHT
Number analyzed (Participants) | 310
Participants | 112

5. Secondary Outcome: Patients Continuing With GANfort® After 18 Weeks
Description: Patients continuing with GANfort® after 18 weeks was assessed as Yes or No.
Time Frame: 18 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Number; unit: Participants
Arm/Group | POAG or OHT
Number analyzed (Participants) | 355
Participants | 329

ADVERSE EVENTS:
Arm/Group | POAG or OHT
Serious Adverse Events (participants affected / at risk) | 1/392
Other Adverse Events (participants affected / at risk) | 0/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POAG or OHT (N=392)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.